CLINICAL TRIAL: NCT02628093
Title: A Randomized Controlled Trial Comparing THUNDERBEAT to the Ligasure Energy Device During Laparoscopic Colon Surgery
Brief Title: A ProspectiveTrial Comparing THUNDERBEAT to the Ligasure Energy Device During Laparoscopic Colon Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1403014955
Record Dates: First submitted 2015-12-04; First posted 2015-12-11 (Estimated); Results first posted 2020-02-06 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- THUNDERBEAT (Other): THUNDERBEAT energy device ( Olympus) will be used for dissection of tissue and ligation of vessels
  Interventions: Device: THUNDERBEAT
- LIGASURE (Other): LIGASURE energy device will be used for dissection of tissue and ligation of vessels
  Interventions: Device: LIGASURE

INTERVENTIONS:
Device: THUNDERBEAT — Tissue dissection and vessels ligation
  Arms: THUNDERBEAT
Device: LIGASURE — Tissue dissection and vessels ligation
  Arms: LIGASURE

SUMMARY:
Prospective randomized controlled study, at Colon and Rectal Surgery, WMC/NYPH. Subjects undergoing Laparoscopic Left Colectomy will be randomized into 1 of 2 groups based on the instrument used for tissue dissection and vessel ligation: Group 1 - THUNDERBEAT Group 2

- Ligasure Population

DETAILED DESCRIPTION:
Prospective randomized controlled study, at Colon and Rectal Surgery, WMC/NYPH. Subjects undergoing Laparoscopic Left Colectomy will be randomized into 1 of 2 groups based on the instrument used for tissue dissection and vessel ligation: Group 1 - THUNDERBEAT Group 2

- Ligasure Population: 60 subjects, with colon neoplasm or diverticulitis will be invited in the study after surgery is deemed necessary Study Procedures: This project will consist only of prospective data collection. No interventions will be done for research purpose. Data will be collected prospectively on: -Patients (before, during and after surgery) -The THUNDERBEAT and LigaSure instruments Data will be collected on data collection sheets and entered in a password protected database Primary Outcomes/Definitions- Overall time for dissection of the soft tissues necessary for specimen removal during colon resection, measured in minutes, from the start of colon mobilization to specimen removal from the abdominal cavity.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will be undergoing a Left Laparoscopic Colon Resection
* Older than 18 years old
* ASA 1 to 3
* Elective surgeries
* Patients who willingly provide informed consent

Exclusion Criteria:

* Morbidly obese patients (BMI >35)
* Patients with acute diverticulitis
* Patients with multiple previous abdominal surgeries
* Patients on anticoagulants
* Patients who can not, tolerate a major surgery
* Patients for whom electrosurgery is contraindicated
* Patients who are pregnant
* Patient with IBDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Milsom, MD, Principal Investigator — WCMC
Locations (1):
- Weill Cornell Medical Center- NYPH, New York, New York, United States

REFERENCES:
- [Derived] Milsom JW, Trencheva K, Momose K, Peev MP, Christos P, Shukla PJ, Garrett K. A pilot randomized controlled trial comparing THUNDERBEAT to the Maryland LigaSure energy device in laparoscopic left colon surgery. Surg Endosc. 2022 Jun;36(6):4265-4274. doi: 10.1007/s00464-021-08765-8. Epub 2021 Nov 1. PMID 34724584

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 73 subjects were enrolled, and 60 of them were randomized into the two groups.
Period: Overall Study
Arm/Group | THUNDERBEAT | LIGASURE
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | THUNDERBEAT | LIGASURE | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Median (Full Range); unit: years] | 54 [31 to 92] | 63 [29 to 88] | 59.5 [29 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 17 | 12 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
Body mass index(BMI) [Mean (Standard Deviation); unit: kgm^2] — BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared.
  kgm^2 | 26.3 (4.3) | 26.4 (4) | 26.3 (4.2)
ASA Class [Median (Full Range); unit: scores on a scale] — American Society of Anesthesiologists Classification (ASA Class) and has 6 levels plus an indicator "E" for an emergency cases.ASA 1: A normal healthy patient, ASA 2: A patient with a mild systemic disease,ASA 3: A patient with a severe systemic disease that is not life-threatening, to ASA 6: A brain-dead patient whose organs are being removed with the intention of transplanting them into another patient.This trial enrolled patients with ASA 1 to 3.
  scores on a scale | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Overall Time for Dissection of the Soft Tissues
Description: from the start of colon mobilization to specimen removal from the abdominal cavity
Time Frame: Day 0 Surgical procedure
Measure: Median (Full Range); unit: minutes
Arm/Group | THUNDERBEAT | LIGASURE
Number analyzed (Participants) | 31 | 29
minutes | 91 [41 to 172] | 77 [38 to 175]
Statistical Analysis 1: Comparison: THUNDERBEAT vs LIGASURE; Because this was a pilot (exploratory) randomized study, no formal sample size calculation was required. Demographic, preoperative, and postoperative variables and the primary outcome were compared between groups (THUNDERBEAT and LigaSure) by the Wilcoxon rank-sum test for continuous variables and the chi-square test/Fisher's exact test for categorical variables, as appropriate. All p-values are two-sided with statistical significance evaluated at the 0.05 alpha level; Test type: Other — Because this was a pilot (exploratory) randomized study, no formal sample size calculation was required; p = 0.214, Wilcoxon (Mann-Whitney) — P value threshold <0.05

2. Primary Outcome: Versatility Score
Description: Total/Composite score (composite of 5 variables:hemostasis;sealing;cutting;dissection;and tissue manipulation) was measured by a score system from 1 to 5 (1 being worst and 5 best) for each of the 5 variables,weighted by Coefficient of Importance with weight distribution as follow: hemostasis 0.275, sealing 0.275, cutting 0.2, dissection 0.15, and tissue Manipulation 0.1.). The final reported score is a weighted average.
Time Frame: Day 0 Surgical procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THUNDERBEAT | LIGASURE
Number analyzed (Participants) | 31 | 29
score on a scale | 4.8 (0.18) | 4.7 (0.22)
Statistical Analysis 1: Comparison: THUNDERBEAT vs LIGASURE; compared between groups by the Wilcoxon rank-sum test; Test type: Other; p = 0.007, Wilcoxon (Mann-Whitney) — P value threshold <0.05

3. Secondary Outcome: Length of Post Surgical Stay in the Hospital
Description: Length of post surgical stay in the hospital measured in days
Time Frame: from Surgery date to the discharge date from the hospital up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | THUNDERBEAT | LIGASURE
Number analyzed (Participants) | 31 | 29
days | 4.5 (3.1) | 5.3 (3.9)

4. Secondary Outcome: Dryness of the Surgical Field Average Score Mean/sd
Description: Measured by score from 1 to 5 where 1 means Heavy bleeding , hemostasis achieved with the instrument with more than 2 attempts, and 5 means No oozing at vessel or tissue site in entire surgical field .
Time Frame: Day 0 Surgical Procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THUNDERBEAT | LIGASURE
Number analyzed (Participants) | 31 | 29
score on a scale | 4.5 (0.38) | 4.4 (0.33)

5. Secondary Outcome: Intraoperative Complication Related to the Energy Devices
Description: Intraoperative adverse event occurrences during surgery due to the energy devices (THUNDERBEAT and LigaSure) measured as categorical variable "Yes" or "No"
Time Frame: Day 0 Surgical procedure
Measure: Number; unit: percentage of total in the group
Arm/Group | THUNDERBEAT | LIGASURE
Number analyzed (Participants) | 31 | 29
percentage of total in the group | 0 | 0

6. Secondary Outcome: Delayed Thermal Injuries Related to Energy Devices
Description: Delayed thermal injuries related to Energy devices that occur after surgery within 30 days of the surgical date, measured as categorical variables "Yes" or "No".
Time Frame: DAY 1 to DAY 30 Postsurgery
Measure: Number; unit: percentage of total number in the group
Arm/Group | THUNDERBEAT | LIGASURE
Number analyzed (Participants) | 31 | 29
percentage of total number in the group | 0 | 0
Statistical Analysis 1: Comparison: THUNDERBEAT vs LIGASURE; Test type: Other; p = 1.0, Fisher Exact — P value threshold <0.05

7. Secondary Outcome: Operative Procedure Time
Description: operative procedure time measured in minutes from the start of the incision to the last stitch in the closure of the surgical incision
Time Frame: Day 0 Surgical Procedure
Measure: Median (Full Range); unit: minutes
Arm/Group | THUNDERBEAT | LIGASURE
Number analyzed (Participants) | 31 | 29
minutes | 176 [113 to 270] | 170 [98 to 265]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Since this is a standard of care procedures no adverse events were recorded. However all intraoperative and postoperative complications were documented as described in the protocol. All the complications that were collected are not qualifying as serous adverse event per protocol.
Arm/Group | THUNDERBEAT | LIGASURE
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 3/31 | 9/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | THUNDERBEAT (N=31) | LIGASURE (N=29)
Postoperative Rectal Bleeding (Injury, poisoning and procedural complications) | 3 | 4
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 2
Wound hematoma incision (Injury, poisoning and procedural complications) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT02628093/Prot_SAP_000.pdf